CLINICAL TRIAL: NCT00263393
Title: Evaluation of a Primary Health Care Intervention for the Prevention of Cardiovascular Disease in Rural Andhra Pradesh
Brief Title: Rural Andhra Pradesh Cardiovascular Prevention Study (RAPCAPS)
Acronym: RAPCAPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Byrraju Foundation (Other); The Future Forum, UK (Unknown)
Responsible Party: Principal Investigator, Dr Rohina Joshi, Research Fellow, The George Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: GI-CA-RAP-A
Record Dates: First submitted 2005-12-06; First posted 2005-12-08 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Myocardial Infarction; Angina Pectoris; Cerebrovascular Accidents; Diabetes Mellitus
Keywords: Myocardial Infarction; Angina Pectoris; Cerebrovascular Accident; Diabetes Mellitus; Cluster randomized design; Community-based intervention trial; Primary Healthcare intervention; Lifestyle advice
MeSH Terms: conditions — Myocardial Infarction; Angina Pectoris; Stroke; Diabetes Mellitus | interventions — Atenolol; Hydrochlorothiazide; Angiotensin-Converting Enzyme Inhibitors; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Health Promotion

ARMS (2):
- Algorithm-based care (Other): An algorithm based approach to increase the identification of high-risk individuals in the community through encouraging opportunistic screening, and to increase the use of appropriate evidence based prevention strategies.
  Interventions: Drug: ASA, Atenolol, hydrochlorothiazide, ACE inhibitor, Statin
- Health-promotion (Other): The health promotion arm has been designed to increase knowledge of the causes of cardiovascular disease and enhance use of preventive behaviours in the general population
  Interventions: Behavioral: Health Promotion

INTERVENTIONS:
Drug: ASA, Atenolol, hydrochlorothiazide, ACE inhibitor, Statin — The first intervention was a clinical algorithm designed to enhance the identification and treatment of high-risk individuals compared to continued usual care. The algorithm was designed to be used by either physician or non-physician health care workers.
  Arms: Algorithm-based care
Behavioral: Health Promotion — The second intervention was a health promotion program designed to increase knowledge of cardiovascular risk factors compared to continued usual practices.
  Arms: Health-promotion

SUMMARY:
This study will evaluate the effectiveness of a novel cardiovascular disease prevention program designed for delivery through existing primary health care services in rural villages in Andhra Pradesh.

The primary aim is to increase the number of high-risk individuals in the population that are appropriately managed with proven, low-cost preventive interventions. The corresponding null hypothesis is therefore that the prevention program will result in no change in the proportion of high-risk individuals identified and treated in villages assigned to intervention compared with those villages assigned to control.

DETAILED DESCRIPTION:
STUDY TYPE This project is a community intervention study that will use a large-scale, cluster-randomised design to compare the management of individuals at high cardiovascular risk in villages assigned to receive the cardiovascular prevention program (intervention) and villages assigned to continue usual practices (control). The definition of high-risk for treatment is based on an established history of previous vascular disease -heart attack or stroke- known hypertension or systolic blood pressure > 160mmHg, or the presence of other risk factors such as smoking, high blood pressure, obesity, older age and family history which combined would result in a very high level of risk.

INTERVENTION PROGRAM TO BE EVALUATED The program to be evaluated comprises: (1) simple strategies designed to facilitate the opportunistic identification of high-risk individuals, (2) clinical algorithms for the implementation of proven preventive interventions based on World Health Organisation recommendations (3) a health promotion campaign designed to aid self-identification and self-referral of high-risk people and (4) simple, structured education programs to assist patients to comply with their treatment.

DATA COLLECTION Data to be collected will comprise an interviewer administered questionnaire with demographic details, basic medical history, cardiovascular risk factors, previous cardiovascular disease and any current treatments. This will be followed by a brief physical examination including measurement of blood pressure, heart rate, weight, height, waist and hip circumferences. Urine will be tested using a dipstick in all and all will have a fasting blood glucose assay. Fasting venous blood samples will be collected for assay of cholesterol, glucose and creatinine from a sample of 1,000.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 years and above
* Personal history of heart attack or stroke
* Presence of other cardiovascular risk factors such as smoking, overweight, diabetes

Exclusion Criteria:

* Mental disability
* Not living in the Study area

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3712 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The proportion of high-risk individuals that have been assessed for cardiovascular risk | 12 months after intevention
The proportion of individuals with correct knowledge about the effects of behavioural determinants of the risk of cardiovascular disease | 12 months from intervention

SECONDARY OUTCOMES:
The proportion of high risk individuals treated with two or more of the recommended drug therapies | 12 months
The knowledge, attitudes and practices of the population about preventable conditions and actions taken to prevent non-communicable disease | 12 months from intervention
The risk factor levels of the population identified as high risk. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce C Neal, Principal Investigator — The George Institute
Locations (1):
- Byrraju Foundation Primary Healthcare Centres in rural West Godavari and East Godavari Dstricts, Bhimavaram, Andhra Pradesh, India

REFERENCES:
- [Background] Chow CK, Joshi R, Gottumukkala AK, Raju K, Raju R, Reddy S, Macmahon S, Neal B. Rationale and design of the Rural Andhra Pradesh Cardiovascular Prevention Study (RAPCAPS): a factorial, cluster-randomized trial of 2 practical cardiovascular disease prevention strategies developed for rural Andhra Pradesh, India. Am Heart J. 2009 Sep;158(3):349-55. doi: 10.1016/j.ahj.2009.05.034. Epub 2009 Jul 15. PMID 19699856
- [Result] Joshi R, Chow CK, Raju PK, Raju KR, Gottumukkala AK, Reddy KS, Macmahon S, Heritier S, Li Q, Dandona R, Neal B. The Rural Andhra Pradesh Cardiovascular Prevention Study (RAPCAPS): a cluster randomized trial. J Am Coll Cardiol. 2012 Mar 27;59(13):1188-96. doi: 10.1016/j.jacc.2011.10.901. No abstract available. PMID 22440219